CLINICAL TRIAL: NCT04257825
Title: The Chili + OURA Sleep Study
Brief Title: Use of Temperature Controlling Mattress Pad for Sleep Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ProofPilot (Industry)
Collaborators: Kryo Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2206
Record Dates: First submitted 2020-01-25; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: In the four week study, participants were randomized into multiple arms, and asked to not use their device for 1 week, and then use it the next. Arms alternated back and forth.
Masking Description: There was no masking in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Off (Other): Individuals were asked to not use their device on weeks 1 and 3 of the study. They were asked to use their device on weeks 2 and 4.
  Interventions: Device: Chili Sleep System
- Initial On (Other): Individuals were asked to not use their device on weeks 2 and 4 of the study. They were asked to use their device on weeks 1 and 3.
  Interventions: Device: Chili Sleep System

INTERVENTIONS:
Device: Chili Sleep System — A mattress pad that cools or warms bed to maintain a constant temperature.

SUMMARY:
A dual arm interventional study in which chliipad and ooler sleep system users voluntarily opt out of using their device for 2 out of 4 weeks. Assessments of sleep via self report and Oura Ring sleep quality and duration.

ELIGIBILITY:
Inclusion Criteria:

* has a chili sleep system
* has an Oura Ring

Exclusion Criteria:

* medically treatable issue
* recent injury
* expected significant travel over study period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Deep Sleep as Measured by Oura Ring | From week 1 to week 2
  Oura Ring is a connected health device worn on the finger that measures sleep. Deep sleep summaries per day will be compared between week 1 and week 2.
Change in self-reported sleep quality via Jenkins Sleep Scale | From week 1 to week 2
  A 8 item self-assessment questionnaire of sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Virtual Study: https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to make data available to other researchers.